CLINICAL TRIAL: NCT05077891
Title: Relationship Between Patient Reported Postpartum Quality of Recovery and Maternal Satisfaction After Cesarean Delivery: A Prospective Observational Study
Brief Title: Postpartum Quality of Recovery & Maternal Satisfaction After C/S
Acronym: QuReS
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Director of Research, University of British Columbia
Other Study IDs: H21-01082
Record Dates: First submitted 2021-09-30; First posted 2021-10-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Measuring patient-oriented outcomes and satisfaction is important to guide meaningful changes in obstetric anesthesia care. Quality of Recovery (QoR) scores are patient rated measures, which provide a global measure of recovery after surgery. They go beyond the measure of physiological variables to include, physical, cognitive, emotive and functional outcomes. Satisfaction, in addition to QoR scores after anaesthesia is an important quality marker. Measuring satisfaction after the birth of a child is a complex and emotive subject. Understanding the factors that can influence maternal satisfaction may improve patient-centred care. Studies have shown that despite favorable clinical outcomes, many women undergoing caesarean deliveries continue to have poor experience with anaesthesia. These poor experiences go beyond inadequate pain control; many are due to poor communication with clinicians, lack of involvement in decision making, lack of provision of high quality education and information and a feeling of inadequate choice and control relating to decisions of the birth of their babies. In non-obstetric studies, satisfaction after anaesthesia has consistently been shown to be dependent on the information patient has received along with the quality of the communication and the quality of the anaesthetist-patient relationship.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speaker
* Older than 19 years of age
* Received a cesarean delivery
* Received a cesarean delivery 24-48 hours prior to time of recruitment

Exclusion Criteria:

* Non-English speaker
* Below the age of 19 years
* Did not receive a cesarean delivery
* Received a cesarean delivery more than 48hrs after time of recruitment

Min Age: 19 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All women above the age of 19 years old whom underwent a caesarean section will be eligible to participate. Women will be surveyed at 24 hours after their cesarean section. Data will be collected by means of validated paper questionnaires administered in person by a study investigator that is not part of clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery Score (ObsQoR-11) | 5 Minutes
  Quality of recovery will be measured using the obstetric quality of recovery score (ObsQoR-11). This is a 11-item, multidimensional recovery scoring tool, which has been validated in this population
Maternal Satisfaction Scale for Cesarean Section (MSSCS) | 5 Minutes
  This 22 item questionnaire measures satisfaction with the anaesthetic, needle insertion, side effects and the theatre atmosphere. Items are rated on a 7-point likert scale from strongly disagree to strongly agree.
Satisfaction with Received Care | 1 Minute
  First open ended question assessing: "What aspects of your care were you most satisfied with?"
Dissatisfaction with Received Care | 1 Minute
  Second open ended question assessing: "What aspects of your care were you most dissatisfied with?"
Improvement of Satisfaction | 1 Minute
  Third and last open ended question assessing: "Do you have any suggestions on what would improve your satisfaction?"

SECONDARY OUTCOMES:
Obstetric History: Gravidity and Preterm | 1 Minute
  Total frequency of gravidity and preterm
Patient Age | 1 Minute
  Patient age in years
Gestational Age | 1 Minute
  Gestational age in total weeks and days
Patient Height | 1 Minute
  Patient height measured in centimeters
Patient Weight | 1 Minute
  Patient weight measured in kilograms
Outcome of Delivery | 1 Minute
  Result of singleton, twins, or other
Neonatal APGARs | 1 Minute
  APGAR scores at 1 minute and minutes
Neonatal Birthweight | 1 Minute
  Neonatal birthweight measured in grams
Patient ASA Status | 1 Minute
  American Society of Anesthesiologists (ASA) physical status classification system ranging from 1 to 6
Pregnancy Medical Conditions | 1 Minute
  Including: pregnancy induced HTN, pre-eclampsia, gestational diabetes, anemia, hyperemesis, cholestasis, and other.
Medical Conditions Outside Pregnancy | 1 Minute
  Including any medical conditions that do not constitute a pregnancy medical condition
Neuraxial Lidocaine | 1 Minute
  Neuraxial agents and dosage administered prior and during the cesarean section procedure.
Neuraxial Bupivicaine | 1 Minute
  dosage administered prior and during the cesarean section procedure.
Neuraxial Morphine | 1 Minute
  dosage administered prior and during the cesarean section procedure.
Neuraxial Fentanyl | 1 Minute
  dosage administered prior and during the cesarean section procedure.
Intraoperative Anxiolytics | 1 Minute
  Intraoperative anxiolytics drug and dose administered prior and during the cesarean section procedure.
Anesthesia Procedure Start | 1 Minute
  Time in military time format
Urgency of Cesarean Delivery | 1 Minute
  Classified as: scheduled, STAT, P1, or P2
Indication for Cesarean Delivery | 1 Minute
  Reason for cesarean delivery
Labour Onset | 1 Minute
  Indicated as: spontaneous, augmented, or induction of labour
Labour Length | 1 Minute
  Length of hours for both first stage and second stage
Pain Relief During Labour | 1 Minute
  Indicated as: epidural/CSE/DPE, Entonox, M&G, or other
Intraoperative Complications | 1 Minute
  Indicated as: hypotension, shivering, nausea, vomiting, itch, failed neuraxial, or other.
Intraoperative Blood Loss | 1 Minute
  Blood loss measured in milliliters.
Postoperative Complications | 1 Minute
  Any medical complication indicated after the caesarean delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Background] Bowyer A, Jakobsson J, Ljungqvist O, Royse C. A review of the scope and measurement of postoperative quality of recovery. Anaesthesia. 2014 Nov;69(11):1266-78. doi: 10.1111/anae.12730. Epub 2014 Jun 2. PMID 24888412
- [Background] Heidegger T, Saal D, Nubling M. Patient satisfaction with anaesthesia - Part 1: satisfaction as part of outcome - and what satisfies patients. Anaesthesia. 2013 Nov;68(11):1165-72. doi: 10.1111/anae.12347. Epub 2013 Aug 8. PMID 23926924
- [Background] Barnett SF, Alagar RK, Grocott MP, Giannaris S, Dick JR, Moonesinghe SR. Patient-satisfaction measures in anesthesia: qualitative systematic review. Anesthesiology. 2013 Aug;119(2):452-78. doi: 10.1097/ALN.0b013e3182976014. PMID 23669268
- [Background] Camann W. Pain, Pain Relief, Satisfaction and Excellence in Obstetric Anesthesia: A Surprisingly Complex Relationship. Anesth Analg. 2017 Feb;124(2):383-385. doi: 10.1213/ANE.0000000000001676. No abstract available. PMID 28098685
- [Background] Kingsley C, Patel S. Patient-reported outcome measures and patient-reported experience measures. BJA Education. 2017;17(4):137-44.
- [Background] Linda D. Results of the National Maternity Experience Survey 2020 2020 [Available from: https://yourexperience.ie/maternity/national-results/.
- [Background] Porter M, van Teijlingen E, Chi Ying Yip L, Bhattacharya S. Satisfaction with cesarean section: qualitative analysis of open-ended questions in a large postal survey. Birth. 2007 Jun;34(2):148-54. doi: 10.1111/j.1523-536X.2007.00161.x. PMID 17542819
- [Background] Stewart MA. Effective physician-patient communication and health outcomes: a review. CMAJ. 1995 May 1;152(9):1423-33. PMID 7728691
- [Background] Cook K, Loomis C. The Impact of Choice and Control on Women's Childbirth Experiences. J Perinat Educ. 2012 Summer;21(3):158-68. doi: 10.1891/1058-1243.21.3.158. PMID 23730127
- [Background] Brooks H, Sullivan WJ. The importance of patient autonomy at birth. Int J Obstet Anesth. 2002 Jul;11(3):196-203. doi: 10.1054/ijoa.2002.0958. PMID 15321548
- [Background] Morgan PJ, Halpern S, Lo J. The development of a maternal satisfaction scale for caesarean section. Int J Obstet Anesth. 1999 Jul;8(3):165-70. doi: 10.1016/s0959-289x(99)80132-0. PMID 15321139
- [Background] Berning V, Laupheimer M, Nubling M, Heidegger T. Influence of quality of recovery on patient satisfaction with anaesthesia and surgery: a prospective observational cohort study. Anaesthesia. 2017 Sep;72(9):1088-1096. doi: 10.1111/anae.13906. Epub 2017 May 16. PMID 28510285
- [Background] Myles PS, Reeves MD, Anderson H, Weeks AM. Measurement of quality of recovery in 5672 patients after anaesthesia and surgery. Anaesth Intensive Care. 2000 Jun;28(3):276-80. doi: 10.1177/0310057X0002800304. PMID 10853209
- [Background] Ciechanowicz S, Howle R, Heppolette C, Nakhjavani B, Carvalho B, Sultan P. Evaluation of the Obstetric Quality-of-Recovery score (ObsQoR-11) following non-elective caesarean delivery. Int J Obstet Anesth. 2019 Aug;39:51-59. doi: 10.1016/j.ijoa.2019.01.010. Epub 2019 Feb 2. PMID 30885691